CLINICAL TRIAL: NCT02969122
Title: Treatment Strategy for Stage IV Gastric Cancer with Positive Peritoneal Cytology As the Only Non-curable Factor (Cy-plus): a Phase 2, Randomized Controlled Trial
Brief Title: Treatment Strategy for Stage IV Gastric Cancer with Positive Peritoneal Cytology As the Only Non-curable Factor
Acronym: Cy-plus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough cases enrolled in the study.
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, President of Peking University Cancer Hospital, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YJZ35
Record Dates: First submitted 2016-11-12; First posted 2016-11-21 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stomach Neoplasm
Keywords: gastric cancer; peritoneal cytology
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy-first (Active Comparator): Patients will receive hyperthermic intraperitoneal chemotherapy (HIPEC) during laparoscopic staging. Then 3 cycles of preoperative chemotherapy and clinical evaluation of chemotherapy will be performed. If the patient's disease is evaluated as progressed, the patient will receive systemic therapy. If it's stable or remission, a second time laparoscopic staging and peritoneal cytology examination will be performed. If peritoneal implant is observed, the patients will receive systemic therapy. If the peritoneal cytology is still positive, the treatment will be decided according to the suggestion of MDT discussion. If the peritoneal cytology is converted negative, standard gastrectomy with D2 lymphadenectomy and extensive intraperitoneal lavage (EIPL) will be performed. Postoperative chemotherapy will be determined according to the pathological evaluation of preoperative chemotherapy response.
  Interventions: Procedure: standard gastrectomy with D2 lymphadenectomy; Procedure: hyperthermic intraperitoneal chemotherapy; Procedure: Extensive intraperitoneal lavage; Other: Preoperative chemotherapy; Other: Postoperative chemotherapy
- Surgery-first (Experimental): Patients in this arm will receive standard gastrectomy with D2 lymphadenectomy after randomization. Hyperthermic intraperitoneal chemotherapy (HIPEC) and extensive intraperitoneal lavage (EIPL) will be applied before abdominal closure. After surgery, 8 cycles of postoperative chemotherapy will be performed.
  Interventions: Procedure: standard gastrectomy with D2 lymphadenectomy; Procedure: hyperthermic intraperitoneal chemotherapy; Procedure: Extensive intraperitoneal lavage; Other: Postoperative chemotherapy

INTERVENTIONS:
Procedure: standard gastrectomy with D2 lymphadenectomy — standard distal or total gastrectomy and accorded D2 lymphadenectomy
Procedure: hyperthermic intraperitoneal chemotherapy — Intraperitoneal docetaxel of 100mg/m2 at 42℃ for 30 minutes
  Other Names: HIPEC
Procedure: Extensive intraperitoneal lavage — Lavage of peritoneal cavity with 1000ml saline for 10 times
  Other Names: EIPL
Other: Preoperative chemotherapy — Oxaliplatin 130mg/m2 D1 S-1 40-60mg Bid D1-14 Repeated every 3 weeks.
  Arms: Chemotherapy-first
Other: Postoperative chemotherapy — SOX regimen postoperative chemotherapy (Oxaliplatin 130mg/m2 D1, S-1 40-60mg Bid D1-14, Repeated every 3 weeks) for surgery-first arm. Regimen for chemotherapy-first arm is determined according to the postoperative pathologic evaluation of response.

SUMMARY:
Gastric cancer with positive is defined as stage IV disease in 7th AJCC/UICC TNM staging system. Controversy exists on the treatment of this part of patients. This trial aimed to explore the optimal treatment strategy for stage IV gastric cancer with positive peritoneal cytology as the only non-curable factor.

DETAILED DESCRIPTION:
In the 7th AJCC/UICC TNM staging system, gastric cancer with positive peritoneal cytology (CY+) is defined as stage IV disease. In NCCN clinical practice guidelines, it is suggested that positive peritoneal cytology in the absence of visible peritoneal implants should be considered as M1 disease and surgery as initial treatment is not recommended for patients with positive peritoneal cytology. However, in the Japanese gastric cancer treatment guidelines 2014, it is suggested that standard gastrectomy can be proposed for patients with no other non-curative factors and if the CY+ status was revealed after surgery, postoperative treatment with S-1 can be recommended as the tentative standard. Previous studies have also proved that extensive intraperitoneal lavage(EIPL) and Hyperthermic Intraperitoneal Chemotherapy(HIPEC) are effective methods for the treatment of peritoneal metastasis.

In order to optimize the treatment strategy of this part of patients, this trial is designed to compare the effectiveness of 2 treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed gastric adenocarcinoma with endoscopic biopsy;
* Pretreatment clinical stage with computed tomography and/or endoscopic ultrasonography;
* Clinical stage cT2-4 N0-3 M0;
* Standard gastrectomy with D2 lymphadenectomy is needed according to the clinicians' evaluation;
* ECOG performance score ≤2, with tolerance of standard gastrectomy and D2 lymphadenectomy;
* Positive peritoneal cytology;
* Signed informed consent.

Exclusion Criteria:

* Remnant gastric cancer, recurrence gastric cancer or multi-primary cancers;
* Intraoperative identified other unresectable factors including other metastasis except positive peritoneal cytology;
* Postoperative pathologically diagnosed as non adenocarcinoma;
* Pregnant or lactate women;
* Child-bearing period adults who refuse to birth control during the trial;
* Uncontrolled epilepsy, CNS disease or mental disorder that may influence the compliance of the patient;
* Severe/active heart disease, including but not limited to acute coronary syndrome, congestive heart failure with less than NYHA II cardiac function, severe arrhythmia that needs drug control, cardiac infarction within 12 month;
* Organ transplantation patients who needs immune suppression therapy;
* Patients who needs emergency surgery because of bleeding, perforation or obstruction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 year

SECONDARY OUTCOMES:
peritoneal recurrence rate | 3 year
Recurrence free survival | 3 year
rate of peritoneal cytology converted to negative | 7 days After the second time laparoscopic staging and peritoneal cytology examination
morbidity and mortality of HIPEC and EIPL | 30 days after HIPEC and EIPL procedures

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Gastrointestinal Cancer Center, Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No